CLINICAL TRIAL: NCT01706081
Title: Acupuncture for Chronic Lymphedema: A Randomized Wait-list Controlled Trial
Brief Title: Acupuncture for Chronic Lymphedema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-210
Record Dates: First submitted 2012-10-10; First posted 2012-10-15 (Estimated); Results first posted 2019-08-29 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2018-04

CONDITIONS: Breast Cancer With Chronic Lymphedema
Keywords: acupuncture
MeSH Terms: interventions — Acupuncture Therapy; Waiting Lists

ARMS (2):
- Acupuncture (Experimental): Patients in the acupuncture group will receive acupuncture treatment twice weekly for six consecutive weeks.
  Interventions: Procedure: Acupuncture
- Wait-list (Experimental): Patients in the wait-list control group will cross over and receive acupuncture twice weekly for 6 consecutive weeks.
  Interventions: Procedure: Wait-list

INTERVENTIONS:
Procedure: Acupuncture — Each treatment will be 30 minutes in duration. Patients will receive two acupuncture treatments each week for six consecutive weeks. Patients will be advised to continue their standard lymphedema treatments such as exercise or use of compression garments if these were in use prior to clinical trial participation.
  Arms: Acupuncture
Procedure: Wait-list — For participants in the wait-list control group, follow-up objective and subjective assessments of lymphedema will be performed after approximately 6 weeks on the wait-list, before onset of acupuncture treatment, following 6 weeks of acupuncture treatment and about 3 months after completion of treatment. BMI will be measured at the same timepoints.
  Arms: Wait-list

SUMMARY:
This study is being done because women have arm swelling for more than 6 months despite wrapping and other treatments. This swelling is called lymphedema. It is the back up of lymph system fluid that causes swelling in the arm. The swelling can just happen, but more commonly it is caused when lymph nodes are removed during cancer surgery. It can develop right after breast cancer treatment or weeks, months or even years later. In our preliminary research, the investigators found that more than 1/3 of the 33 patients showed at least a 30% reduction in lymphedema following acupuncture treatment and there were no serious adverse events during the treatment or 6 month followup.

This study will include a larger group of patients. Patients will be assigned to one of two groups, and results of the groups will be compared to see if acupuncture can reduce lymphedema and whether the effect lasts after acupuncture treatment is completed.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18 or older
* Lymphedema in an arm as a result of surgery, chemotherapy, and/or radiation therapy for breast cancer per breast surgeon or medical oncologist
* Patients must have received a clinical diagnosis of lymphedema for at least 6 months and no more than 5 years. This timeframe allows ample time for any surgically related non lymphedema swelling to subside by 6 months post-surgery, while a cap of 5 years will capture the broadest range of cases, and has been used as a timeframe in several studies including our pilot study.
* The affected arm must be >2cm larger than the unaffected arm. Differences of 2 cm or more between the affected and unaffected arm are considered by experts to be clinically significant. Each affected arm will be measured in two areas: upper arm and forearm.

The larger of the two measures-upper arm or forearm- will be used for analysis.

* Classified as International Society of Lymphology (ISL) stage II or higher as determined by an MSKCC Certified Lymphedema Therapist (CLT).

Exclusion Criteria:

* Bilateral lymphedema
* Previous acupuncture treatment for lymphedema
* Concurrent diuretic use
* History of primary (congenital) lymphedema
* Pregnant or planning to become pregnant during the course of the study
* Has an implanted electronically charged medical device

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-10; Primary Completion 2018-04-11 (Actual); Study Completion 2018-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ting Bao, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acupuncture | Wait-list
Started | 40 | 42
Completed | 40 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acupuncture | Wait-list | Total
Number analyzed (Participants) | 40 | 42 | 82
Age, Continuous [Median (Full Range); unit: years] | 65 [54 to 71] | 58 [49 to 70] | 61 [49 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 42 | 82
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 31 | 32 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 42 | 82

OUTCOME MEASURES:

1. Primary Outcome: Lymphedema as Measured at Baseline and at 6 Weeks
Description: Changes in lymphedema between groups, as measured by mean arm circumference assessed at baseline and after 6 weeks from baseline.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Acupuncture | Wait-list
Number analyzed (Participants) | 40 | 42
cm
  Baseline | 4.74 (2.23) | 4.82 (2.32)
  6 weeks | 4.29 (2.67) | 4.76 (2.68)

2. Secondary Outcome: Measurements for Bioimpedance for Treatment Arms at Baseline and 6 Weeks
Description: Bioimpedance measured using Impedimed L-Dex U400, which measures the rate of electrical current transmission through tissues and estimate fluid content in a lymphedematous limb compared with the normal limb.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: ohms
Arm/Group | Acupuncture | Wait-list
Number analyzed (Participants) | 40 | 42
ohms
  Baseline | 38.6 (30.4) | 42.2 (32.3)
  6 Week | 35.9 (27.4) | 40.3 (35.6)

3. Secondary Outcome: Number of Participants Evaluated for Adverse Events
Time Frame: 1. 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Wait-list
Number analyzed (Participants) | 40 | 42
Participants | 40 | 42

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Acupuncture | Wait-list
All-Cause Mortality (participants affected / at risk) | 6/40 | 7/42
Serious Adverse Events (participants affected / at risk) | 12/40 | 7/42
Other Adverse Events (participants affected / at risk) | 20/40 | 11/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acupuncture (N=40) | Wait-list (N=42)
Anemia (Blood and lymphatic system disorders) | 2 | 0
Gastric Hemorrhage (Gastrointestinal disorders) | 1 | 0
Gen disorders & admin site conditions Other, spec (General disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin & subcutaneous tissue disorders Other, spec (Skin and subcutaneous tissue disorders) | 1 | 2
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Acupuncture (N=40) | Wait-list (N=42)
Anemia (Blood and lymphatic system disorders) | 3 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 3
Lymphocyte count decreased (Investigations) | 2 | 1
Neutrophil count decreased (Investigations) | 4 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Platelet count decreased (Investigations) | 2 | 0
White blood cell decreased (Investigations) | 4 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-29): https://cdn.clinicaltrials.gov/large-docs/81/NCT01706081/Prot_SAP_000.pdf